CLINICAL TRIAL: NCT05852587
Title: Xylitol Use for Decolonization of C. Difficile in Patients With Inflammatory Bowel Disease
Brief Title: Xylitol Use for Decolonization of C. Difficile in Patients With IBD
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jessica Ravikoff Allegretti, Director, Crohn's and Colitis Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023P001327
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Inflammatory Bowel Diseases; Clostridioides Difficile Infection
Keywords: Crohn's Disease; Ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Clostridium Infections; Crohn Disease; Colitis, Ulcerative | interventions — Xylitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose A of Xylitol (Experimental): Patients in this arm will be receiving 7.5g/day of Xylitol over a 4 week period.
  Interventions: Drug: Xylitol
- Dose B of Xylitol (Experimental): Patients in this are will be receiving 15g/day of Xylitol over a 4 week period.
  Interventions: Drug: Xylitol
- Placebo (Placebo Comparator): Patients in this arm will be receiving placebo over a 4 week period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xylitol — Xylitol is a sugar alcohol and considered a GRAS substance by the FDA. Xylitol is also an FDA approved as a food additive. Xylitol will be used as a treatment for the decolonization of C. difficile and will be given in gel capsules. The xylitol provided will be prepared by the BWH investigational drug service and ordered from MEDISCA suppliers. It will be 100% pure. Xylitol has a distinct taste and therefore it will be administered in gel capsules as opposed to an oral solution to maintain blinding.
  Arms: Dose A of Xylitol; Dose B of Xylitol
Drug: Placebo — The placebo will be administered by the BWH investigational drug services. The placebo will be composed of cellulose microcrystal.
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, dose-ranging study to assess the safety and efficacy of xylitol as an oral therapeutic for decolonization of C. difficile in IBD patients. A total of 99 patients who meet eligibility criteria will be randomized 1:1:1 to one of two xylitol doses or placebo arm. All arms will receive an identical capsule dosing for four weeks. Microbiome assessment and C. difficile testing will be performed at baseline, week 4, 8, 26, and 52.

DETAILED DESCRIPTION:
This randomized placebo-controlled dose-finding trial will assess the safety and efficacy of xylitol as an oral therapeutic for decolonization of C. difficile in the IBD patient population.

Participants with confirmed IBD diagnosis who are scheduled for an outpatient colonoscopy for any reason at Brigham and Women's Hospital or clinic appointment at the Crohn's and Colitis Center will be eligible for screening. Participants will be screened for C. difficile colonization via colonic wash sampling during colonoscopy or whole stool following a clinic appointment.

Participants may only have inactive or mild IBD based in clinical scores (see inclusion criteria) to be eligible for screening. Risk factors for colonization will be assessed by comparing colonized vs. not colonized patients.

Participants who are found to be colonized will be randomized 1:1:1 to either placebo or one of two dosing groups of xylitol. The dose A treatment arm will receive 7.5 grams daily of xylitol via gel capsule for 4 weeks. The dose B treatment arm will receive 15 grams daily of xylitol via gel capsule for 4 weeks. The placebo arm will receive identical capsule dosing for 4 weeks. Participants will end dosing at week 4, but monitoring will continue through week 52. Both participants and study team will be blinded to treatment arm allocation.

The primary endpoints assessed are decolonization at week 8 as well as safety and tolerability through week 8. In addition, secondary efficacy outcomes including IBD disease activity and development of CDI, which will be evaluated at week 8, week 26 and week 52. Disease activity and symptoms will be recorded from informed consent through the week 52 trial visit.

Stool samples for biomarker assessments and C. difficile testing will be collected at scheduled trial visits per Schedule of Assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Male or female ≥ 18 years of age
3. IBD diagnosis (CD, UC or indeterminant Colitis will be permitted)
4. Inactive or mild IBD (HBI score ≤ 7; Partial Mayo score ≤ 4)
5. Presenting for outpatient colonoscopy or clinic appointment for any indication

Exclusion Criteria:

1. Unable to provide consent
2. Patients with previous colectomy, ostomy, J-pouch, or previous colon surgery (excluding appendectomy)
3. Unable to complete study procedures
4. Chronic use of antibiotics
5. Inability or unwillingness to swallow capsules
6. Allergy to xylitol
7. Stool positive for Listeria monocytogenes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2032-01-01 (Estimated); Study Completion 2033-01-01 (Estimated)

PRIMARY OUTCOMES:
C.difficile decolonization | 8 weeks
  Absence of C. difficile via PCR in week 8 stool sample
safety and tolerability | 8 weeks
  Subject incidence of treatment-emergent adverse events (including treatment-emergent adverse events for clinically significant changes in laboratory parameters and vital signs)

SECONDARY OUTCOMES:
biomass of C.difficile | 8 weeks
  Change in biomass of C. difficile
IBD clinical outcomes | 8 weeks
  Clinical Remission: Partial Mayo score less than 1 & HBI score less than 5 Clinical Response: A decrease from baseline in the HBI score or SCCAI score by three points
IBD clinical outcomes | 52 weeks
  Clinical Remission: Partial Mayo score less than 1 & HBI score less than 5 Clinical Response: A decrease from baseline in the HBI score or SCCAI score by three points
C. difficile infection | 52 weeks
  Incidence of patients developing CDI

CONTACTS AND LOCATIONS:
Overall Officials: Jessica R Allegretti, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No